CLINICAL TRIAL: NCT03538340
Title: Randomized, Single-Blinded, Controlled Trial Using Intraoperative Cryoanalgesia for Extended Pain Management Following Thoracotomy: ICE Study
Brief Title: Intraoperative Cryoanalgesia for Extended Pain Management Following Thoracotomy
Acronym: ICE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: AtriCure, Inc. (Industry)
Responsible Party: Principal Investigator, Joseph S. Friedberg, MD, Professor; Surgeon-in-Chief, UMMS Division of Thoracic Surgery, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HP-00079115
Record Dates: First submitted 2018-03-07; First posted 2018-05-29 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Chronic Post-thoracotomy Pain; Acute Post-thoracotomy Pain; Post-thoracotomy Pain Syndrome
Keywords: Thoracotomy; Cryoanalgesia; Pain
MeSH Terms: conditions — Pain | interventions — Tea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control Arm (Active Comparator): Control Arm: Surgery without intercostal Cryoanalgesia + Standard of Care (thoracic epidural)
  Interventions: Procedure: Thoracic Epidural
- Study Arm (Experimental): Study Arm: Surgery with intercostal Cryoanalgesia + Standard of Care (thoracic epidural)
  Interventions: Procedure: Thoracic Epidural; Procedure: Intercostal Cryoanalgesia

INTERVENTIONS:
Procedure: Thoracic Epidural — The control arm will receive standard of care pain management which includes a Thoracic Patient Controlled Epidural
Procedure: Intercostal Cryoanalgesia — The study arm will receive standard of care pain management which includes a Thoracic Epidural plus Intraoperative Intercostal Cryoanalgesia
  Arms: Study Arm

SUMMARY:
The ICE Study study will compare standard therapy (thoracic epidural) versus a novel approach (Cryoanalgesia combined with thoracic epidural) in subjects undergoing unilateral thoracotomy.

DETAILED DESCRIPTION:
The ICE Study is a single institution pilot study designed to compare standard therapy (i.e., thoracic epidural) versus a novel approach (i.e., Cryoanalgesia combined with thoracic epidural) to address the need for better management of acute and long-term pain in the general thoracic surgery patient population. The study's primary objective will be to demonstrate if the new intraoperative pain management approach [i.e., intercostal Cryoanalgesia in conjunction with thoracic epidural] provides superior short-term and long-term analgesia efficacy in patients undergoing unilateral thoracotomy as compared to the current institutional standard of care (i.e., thoracic epidural). Patients will be randomized in a 1:1 design.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing unilateral thoracotomy for non-cardiac surgery
* Age 18-85 years of age; male or female
* Acceptable surgical candidate including use of general anesthesia
* Willing and able to provide written informed consent
* Willing and able to return for scheduled follow-up visits

Exclusion Criteria:

* Prior major surgery within the last 6-months
* Documented psychiatric disease
* Documented chronic pain syndrome
* Current use of prescription opioids
* Documented history of substance abuse
* Functional disability or impairment (ECOG score = 0 or 1)
* Current pregnancy
* Patients currently enrolled in another research study that could directly affect results of either study
* Physical or mental condition that would interfere with patient's self-assessment of pain
* A medical condition that in the investigator's opinion could adversely impact the patient's participation or safety, conduct of the study or interferes with the pain assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Total narcotic use post-thoracotomy. | 6 months
  The primary outcome measure of this study is to determine if the addition of Cryoanalgesia to standard of care post thoracotomy pain control, results in decreased pain and/or narcotic use at time points ranging from perioperative to six months post discharge.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) Assessment of post-thoracotomy pain | 6 months
  Visual Analog Scale will be used to assess pain levels (0-10 range scale with 0=no pain and 10= worse pain ever
Quality of Life (SF-36) changes from baseline to 6-months | 6 months
  Assessment of the impact of pain on quality of life (questions using varied assessment scales: rating general health from excellent to poor; yes-no; none to very severe; not at all to extremely; all of the time to none of the time; true-false
Allodynia Assessment | 6 months
  Allodynia screening and assessments will assess the levels of skin hypersensitivity associated with neuropathic pain following thoracotomy and will be performed at predetermined time points
Mankoski Pain Scale Assessment of post-thoracotomy pain | 6 months
  Mankoski Pain Scale will be used to assess pain levels (scale ranging from 0 to 10 with 0 = no pain to 10 = worse pain ever

CONTACTS AND LOCATIONS:
Overall Officials: Joseph S Friedberg, MD, Principal Investigator — U Maryland, Baltimore
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No